CLINICAL TRIAL: NCT02736682
Title: Single Dose Ceftriaxone and Metronidazole Versus Multiple Doses for Antibiotic Prophylaxis at Elective Cesarean Section in Mulago Hospital. A Randomized Clinical Trial.
Brief Title: Single Dose Ceftriaxone and Metronidazole Versus Multiple Doses for Antibiotic Prophylaxis at Elective Cesarean Section.
Acronym: SDvMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013/HD07/658U
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Post Operative Infections
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single dose antibiotic (Experimental): 2g of intra venous Ceftriaxone and 500 mgs Intra venous metronidazole is administered to the mothers as a Single dose pre-operative30-60 minutes before surgery.
  Interventions: Drug: Single dose antibiotic
- multiple dose antibiotic. (Active Comparator): Multiple doses of IV Ceftriaxone 1g and metronidazole 500mgs given to the mother during surgery there after Ceftriaxone 1g every day for 3 days and IV metronidazole 500 mgs every 8 hours for 3 days.
  Interventions: Drug: Multiple dose antibiotic

INTERVENTIONS:
Drug: Single dose antibiotic — Single dose arm receive 2g of IV Ceftriaxone and 500 mgs ofIntra venous Metronidazole given to the mothers 30-60 minutes pre operative.
  Other Names: Epicefin, E.I.P.I.CO.Unique Metrogyl injection.
  Arms: Single dose antibiotic
Drug: Multiple dose antibiotic — Multiple dose arm receive 1 g of IV Cetriaxone plus 500 mgs during surgery and there after IV ceftriaxone once a day for 3 days and IV Metronidazole 500mgs during surgery and there after every 8 hours for 3 days.
  Other Names: Epicefin, E.I.P.I.CO, Unique Metrogyl injection
  Arms: multiple dose antibiotic.

SUMMARY:
Delivery by Cesarean section is increasing worldwide and this is the most important risk factor for post partum infection where there is a 5-20% risk of developing post partum infection than women who deliver vaginally Provision of single dose broad spectrum intravenous antibiotics 30-60 minutes before cesarean section has been found to be as effective as multiple doses in reducing post operative infections. At Mulago National referral Hospital mothers who have had elective and are at low risk of post partum infection also receive multiple doses of intravenous antibiotics for up to 7 days. The rationale of the study is to further inform us that single dose preoperative antibiotic prophylaxis is effective in prevention of post operative infection in mothers delivered by elective cesarean section.

DETAILED DESCRIPTION:
This is going to be an open label randomized controlled clinical trial that will involve 174 mothers delivered by elective cesarean section in Mulago National Referral hospital ward 5B antenatal and post natal wards.

Mulago hospital is at the apex of a 6 tier health system and is the largest public hospital with 31,400 deliveries annually 26.14% by cesarean section and of these 5.6% are elective cesarean sections.

Simple randomization was done where 174 cards were numbered 1-174 {(87 labelled Single Dose (SD) and 87 labelled Multiple Dose (MD)} inserted in an envelop shuffled and then the mother was allowed to pick a card randomly. This was done by the research assistant who reviewed the mother again in theater to ascertain if they still met the eligibility before the intervention was done.

Method This will be an open label single center superiority randomized clinical trial involving 174 eligible participants (87 in each arm) who will have delivered by elective cesarean section in Mulago hospital. They will be randomly allocated into two arms. One arm will receive single dose IV ceftriaxone 2g and metronidazole 500mg 30-60 minutes before the operation and the second arm will receive IV ceftraixone 1g with 500 mg of metronidazole during the operation and continue for 72 hours and discharged with oral antibiotics.

The mothers will be reviewed twice daily for evidence of infection. Their vitals (BP, Pulse, Temperature and respiratory rate), state of the wound and uterus, amount color and smell of the lochia during the first 2-3 post operative days. Both arms will have a 14 day follow up where they will come back for review on the 7th and 14th post operative day.

Objective:

The general objective is to compare the incidence of post operative infections among mothers that receive single dose pre operative Ceftriaxone and metronidazole compared to multiple doses at delivery by elective cesarean section in Mulago National Referral Hospital. at 14 day post operative.

ELIGIBILITY:
Inclusion Criteria:

* Antenatal mothers who have an indication for elective cesarean section in New Mulago hospital.

Exclusion Criteria:

* Mothers who have a history of allergy to any of the drugs in the study, Mother with visible infection at any site or elevated body temperature before going to theatre, Those with rapture of membranes, Mothers who went into labor, Mother who has had use of antibiotics in the last 7 days, WHO Clinical HIV stage III and IV and mothers who do not consent to the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Post operative wound infections | 14 days
  Compare for incidence of post operative wound infection among mothers that receive single dose versus multiple dose antibiotics

SECONDARY OUTCOMES:
clinical endometritis | 14 days
  Compare the incidence of clinical endometritis among mothers that receive single versus multiple dose antibiotics
febrile morbidity | 14 days
  compare the incidence of post operative febrile morbidity among mothers that receive single versus multiple doses

CONTACTS AND LOCATIONS:
Overall Officials: Mugisa Alex Gideon, MBChB., Principal Investigator — Makerere University Collage of Health Sciences, Department of Obstetrics and Gynecology; Paul Kiondo, MD, MMeD,PhD, Study Director — Makerere University Collage of Health Sciences, Department of Obstetrics and Gynecology; Imelda Namagembe, MD, MMeD, MPH, Study Director — Mulago NAtional Referral Hospital
Locations (1):
- Mulago National Refferal Hospital, Kampala, Uganda

REFERENCES:
- [Derived] Williams MJ, Carvalho Ribeiro do Valle C, Gyte GM. Different classes of antibiotics given to women routinely for preventing infection at caesarean section. Cochrane Database Syst Rev. 2021 Mar 4;3(3):CD008726. doi: 10.1002/14651858.CD008726.pub3. PMID 33661539